CLINICAL TRIAL: NCT01302834
Title: Phase III Trial of Radiotherapy Plus Cetuximab Versus Chemoradiotherapy in HPV-Associated Oropharynx Cancer
Brief Title: Radiation Therapy With Cisplatin or Cetuximab in Treating Patients With Oropharyngeal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-1016; CDR0000695731; NCI-2011-02638 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Results first posted 2020-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer; Precancerous Condition
Keywords: stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; human papilloma virus infection
MeSH Terms: conditions — Head and Neck Neoplasms; Precancerous Conditions; Squamous Cell Carcinoma of Head and Neck; Papillomavirus Infections | interventions — Cetuximab; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMRT + Cisplatin (Active Comparator): Intensity-modulated radiotherapy (IMRT) with concurrent cisplatin
  Interventions: Drug: cisplatin; Radiation: IMRT
- IMRT + Cetuximab (Active Comparator): Intensity-modulated radiotherapy (IMRT) with concurrent cetuximab
  Interventions: Biological: cetuximab; Radiation: IMRT

INTERVENTIONS:
Biological: cetuximab — 400 mg/m2 IV 5-7 days before IMRT then 250 mg/m2 IV weekly for 7 weeks
  Arms: IMRT + Cetuximab
Drug: cisplatin — 100 mg/m2 IV on days 1 and 22 of IMRT
  Arms: IMRT + Cisplatin
Radiation: IMRT — 35 fractions over 6 weeks, 6 fractions per week, 2 Gray per fraction to total dose of 70 Gy.
  Other Names: intensity-modulated radiotherapy; intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether radiation therapy is more effective with cisplatin or cetuximab in treating oropharyngeal cancer.

PURPOSE: This phase III trial is studying radiation therapy with cisplatin or cetuximab to see how well it works in treating patients with oropharyngeal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether substitution of cisplatin with cetuximab will result in comparable 5-year overall survival.

Secondary

* To monitor and compare progression-free survival for "safety".
* To compare patterns of failure (locoregional vs distant).
* To compare acute toxicity profiles (and overall toxicity burden).
* To compare overall quality of life (QOL) short-term (< 6 months) and long-term (1 year).
* To compare QOL Swallowing Domains short-term and long-term.
* To compare clinician-reported versus patient-reported CTCAE toxicity events.
* To explore differences in the cost effectiveness of cetuximab as compared to cisplatin.
* To explore differences in work status and time to return to work.
* To compare patient-reported changes in hearing.
* To compare CTCAE v. 4 late toxicity at 1, 2, and 5 years.
* To evaluate the effect of tobacco exposure (and other exposures) as measured by standardized computer-assisted self interview (CASI) on overall survival and progression-free survival.
* To pilot CASI collection of patient reported outcomes in a cooperative group setting.
* To determine whether specific molecular profiles are associated with overall or progression-free survival.
* To investigate associations between changes in serum biomarkers or human papilloma virus (HPV)-specific cellular immune responses measured at baseline and three months with overall or progression-free survival.

OUTLINE: This is a multicenter study. Patients are stratified according to T stage (T1-2 vs T 3-4), N stage (N0-2a vs N2b-3), Zubrod performance status (0 vs 1), and smoking history (≤ 10 pack-years vs > 10 pack-years). Patients are randomized to 1 of 2 treatment arms.

Patients may complete quality-of-life questionnaires and risk factors for head and neck cancer surveys at baseline, periodically during study, and at follow-up for 1 year.

After completion of study therapy, patients are followed up at 1-3 months, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically (histologically or cytologically) proven diagnosis of squamous cell carcinoma (including the histological variants papillary squamous cell carcinoma and basaloid squamous cell carcinoma) of the oropharynx (tonsil, base of tongue, soft palate, or oropharyngeal walls).
2. Patients must be positive for p16, determined by central review prior to randomization.
3. Patients must have clinically or radiographically evident measurable disease at the primary site or at nodal stations. Tonsillectomy or local excision of the primary without removal of nodal disease is permitted, as is excision removing gross nodal disease but with intact primary site. Limited neck dissections retrieving ≤ 4 nodes are permitted and considered as non-therapeutic nodal excisions. Fine needle aspirations of the neck are insufficient due to limited tissue for retrospective central review. Biopsy specimens from the primary or nodes measuring at least 3-5 mm are required.
4. Clinical stage T1-2, N2a-N3 or T3-4, any N (AJCC, 7th ed.; see Appendix III), including no distant metastases, based upon the following minimum diagnostic workup:

   * General history and physical examination by a radiation oncologist and medical oncologist within 8 weeks prior to registration;
   * Examination by an ear, nose, and throat (ENT) or head and neck surgeon, including laryngopharyngoscopy (mirror and/or fiberoptic and/or direct procedure) within 8 weeks prior to registration;
   * One of the following combinations of imaging is required within 8 weeks prior to registration:

     1. A computerized tomography (CT) scan of the neck (with contrast) and a chest CT scan (with or without contrast);
     2. or a magnetic resonance imaging (MRI) scan of the neck (with contrast) and a chest CT scan (with or without contrast);
     3. or a CT scan of neck (with contrast) and a positron emission tomography (PET)/CT of neck and chest (with or without contrast);
     4. or an MRI of the neck (with contrast) and a PET/CT of neck and chest (with or without contrast).

   Note: A CT scan of neck and/or a PET/CT performed for radiation planning and read by a radiologist may serve as both staging and planning tools.
5. Zubrod Performance Status 0-1 within 2 weeks prior to registration
6. Age ≥ 18;
7. Complete blood count (CBC)/differential obtained within 2 weeks prior to registration on study, with adequate bone marrow function, defined as follows:

   * Absolute neutrophil count (ANC) > 1,500 cells/mm3;
   * Platelets > 100,000 cells/mm3;
   * Hemoglobin (Hgb) > 8.0 g/dl; Note: The use of transfusion or other intervention to achieve Hgb > 8.0 g/dl is acceptable.
8. Adequate hepatic function, defined as follows:

   * Bilirubin < 2 mg/dl within 2 weeks prior to registration;
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 3 x the upper limit of normal within 2 weeks prior to registration;
9. Adequate renal function, defined as follows:

   • Serum creatinine < 1.5 mg/dl within 2 weeks prior to registration or creatinine clearance (CCr) ≥ 50 ml/min within 2 weeks prior to registration determined by 24-hour collection or estimated by Cockcroft-Gault formula:

   CCr male = [(140 - age) x (wt in kg)] [(Serum Cr mg/dl) x (72)] CCr female = 0.85 x (CCr male)
10. Patients must provide their smoking history (for stratification) via the computer-assisted self interview (CASI) head and neck risk factor survey tool.
11. Negative serum pregnancy test within 2 weeks prior to registration for women of childbearing potential;
12. Women of childbearing potential and male participants must agree to use a medically effective means of birth control throughout their participation in the treatment phase of the study and until at least 60 days following the last study treatment.
13. Patients who are human immunodeficiency virus (HIV) positive but have no prior acquired immune deficiency syndrome (AIDS) -defining illness and have CD4 cells of at least 350/mm3 are eligible. Patient HIV status must be known prior to registration. Patients must not be sero-positive for Hepatitis B (Hepatitis B surface antigen positive or anti-hepatitis B core antigen positive) or sero-positive for Hepatitis C (anti-Hepatitis C antibody positive). However, patients who are immune to hepatitis B (anti-Hepatitis B surface antibody positive) are eligible (e.g. patients immunized against hepatitis B). HIV-positive patients must not have multi-drug resistant HIV infection or other concurrent AIDS-defining conditions.
14. Patient must provide study specific informed consent prior to study entry, including consent for mandatory submission of tissue for required, central p16 review and consent to participate in the computer-assisted self interview (CASI) survey questions regarding smoking history.

Exclusion Criteria:

1. Cancers considered to be from an oral cavity site (oral tongue, floor mouth, alveolar ridge, buccal or lip), nasopharynx, hypopharynx, or larynx, even if p16 positive, are excluded. Carcinoma of the neck of unknown primary site origin (even if p16 positive) are excluded from participation.
2. Stage T1-2, N0-1;
3. Distant metastasis or adenopathy below the clavicles;
4. Gross total excision of both primary and nodal disease; this includes tonsillectomy, local excision of primary site, and nodal excision that removes all clinically and radiographically evident disease.
5. Simultaneous primaries or bilateral tumors;
6. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible);
7. Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable;
8. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields;
9. Severe, active co-morbidity, defined as follows:

   * 9.1 Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
   * 9.2 Transmural myocardial infarction within the last 6 months;
   * 9.3 Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
   * 9.4 Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration;
   * 9.5 Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol.
   * 9.6 Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition with immune compromise greater than that noted in Section 3.1.13; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
10. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
11. Prior allergic reaction to cisplatin or cetuximab;
12. Prior cetuximab or other anti-EGFR therapy.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 987 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2025-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andy M. Trotti, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; Maura Gillison, MD, PhD, Principal Investigator — Ohio State University
Locations (185):
- United States (183):
  - Providence Cancer Center, Anchorage, Alaska
  - Auburn Radiation Oncology, Auburn, California
  - Roy and Patricia Disney Family Cancer Center at Providence Saint Joseph Medical Center, Burbank, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - Enloe Cancer Center at Enloe Medical Center, Chico, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Kaiser Permanente - Division of Research - Oakland, Oakland, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Santa Clara, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Solano Radiation Oncology Center, Vacaville, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - McKee Medical Center, Loveland, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - North Broward Medical Center, Deerfield Beach, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Integrated Community Oncology Network at Southside Cancer Center, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network, Jacksonville Beach, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Integrated Community Oncology Network - Orange Park, Orange Park, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Florida Cancer Center - Palatka, Palatka, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - Flagler Cancer Center, Saint Augustine, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Georgia Cancer Center for Excellence at Grady Memorial Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Parkview Regional Cancer Center at Parkview Health, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen General Hospital, Goshen, Indiana
  - Community Regional Cancer Care at Community Hospital East, Indianapolis, Indiana
  - Community Regional Cancer Care at Community Hospital North, Indianapolis, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - NSMC Cancer Center - Peabody, Danvers, Massachusetts
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Cancer Institute of Cape Girardeau, LLC, Cape Girardeau, Missouri
  - Kansas City Cancer Centers - South, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Barnes-Jewish West County Hospital, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - Billings Clinic - Downtown, Billings, Montana
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Nebraska Medical Center, Omaha, Nebraska
  - Renown Institute for Cancer at Renown Regional Medical Center, Reno, Nevada
  - Payson Center for Cancer Care at Concord Hospital, Concord, New Hampshire
  - Seacoast Cancer Center at Wentworth - Douglass Hospital, Dover, New Hampshire
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Monmouth Medical Center, Long Branch, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Lourdes Regional Cancer Center, Binghamton, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center, Middleburg Heights, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Precision Radiotherapy at University Pointe, West Chester, Ohio
  - UHHS Westlake Medical Center, Westlake, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Dubs Cancer Center at Rogue Valley Medical Center, Medford, Oregon
  - Providence Cancer Center at PMCC, Medford, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - St. Mary Regional Cancer Center, Langhorne, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - Coastal Cancer Center at Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Northwest Cancer Specialists at Vancouver Cancer Center, Vancouver, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - Theda Care Cancer Institute, Appleton, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
- Canada (2):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - McGill Cancer Centre at McGill University, Montreal, Quebec

REFERENCES:
- [Result] Gillison ML, Trotti AM, Harris J, Eisbruch A, Harari PM, Adelstein DJ, Jordan RCK, Zhao W, Sturgis EM, Burtness B, Ridge JA, Ringash J, Galvin J, Yao M, Koyfman SA, Blakaj DM, Razaq MA, Colevas AD, Beitler JJ, Jones CU, Dunlap NE, Seaward SA, Spencer S, Galloway TJ, Phan J, Dignam JJ, Le QT. Radiotherapy plus cetuximab or cisplatin in human papillomavirus-positive oropharyngeal cancer (NRG Oncology RTOG 1016): a randomised, multicentre, non-inferiority trial. Lancet. 2019 Jan 5;393(10166):40-50. doi: 10.1016/S0140-6736(18)32779-X. Epub 2018 Nov 15. PMID 30449625
- [Derived] Gharzai LA, Morris E, Schipper MJ, Kidwell KM, Nguyen-Tan PF, Rosenthal DI, Gillison ML, Jordan RC, Garden AS, Koyfman SA, Caudell JJ, Blakaj DM, Dunlap NE, Krempl GA, Longo JM, Jones CU, Gensheimer MF, Galloway TJ, DeMora L, Le QT, Shah JL, Suresh K, Mierzwa M. Treatment Interruption and Outcomes in Head and Neck Cancer: A Secondary Analysis of 3 Randomized Clinical Trials. JAMA Otolaryngol Head Neck Surg. 2025 Dec 4:e254203. doi: 10.1001/jamaoto.2025.4203. Online ahead of print. PMID 41343184
- [Derived] Quan DL, Grauer JS, Sunkara PR, Cramer JD. Surgical salvage of human papillomavirus-positive oropharyngeal cancer: Secondary analysis of a randomized controlled trial. Cancer. 2023 Feb 1;129(3):376-384. doi: 10.1002/cncr.34562. Epub 2022 Nov 19. PMID 36401615
- [Derived] Psyrri A, Rampias T, Vermorken JB. The current and future impact of human papillomavirus on treatment of squamous cell carcinoma of the head and neck. Ann Oncol. 2014 Nov;25(11):2101-2115. doi: 10.1093/annonc/mdu265. Epub 2014 Jul 23. PMID 25057165
- Available data/document: Individual Participant Data Set: NCT01302834 — https://nctn-data-archive.nci.nih.gov/ — Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sites were required to submit participant tumor tissue for central p16 evaluation within one week of registration. If participants were determined to be p16-positive and continued on the study, then treatment arm was assigned. Of 987 participants registered, 849 were randomized.
Period: Overall Study
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Started | 424 | 425
Eligible (All eligible participants) | 406 | 399
Started Treatment (Eligible and started study treatment) | 398 | 394
AE Assessed 1 Month Post-treatment (PT) (Eligible, started study treatment, and had adverse events (AE) assessment 1 month post-treatment) | 369 | 363
AE Assessed 3 Months PT (Eligible, started study treatment, and had adverse events assessment 3 months post-treatment) | 359 | 367
AE Assessed 6 Months PT (Eligible, started study treatment, and had adverse events assessment 6 months post-treatment) | 361 | 352
AE Assessment 1 Year PT (Eligible, started study treatment, and had adverse events assessment 1 year post-treatment) | 360 | 351
AE Assessed 2 Years PT (Eligible, started study treatment, and had adverse events assessment 2 years post-treatment) | 311 | 303
AE Assessed 5 Years PT (Eligible, started study treatment, and had adverse events assessment 5 years post-treatment) | 92 | 86
Dental Health Assessed 1 Year PT (Eligible, started study treatment, and had dental health assessment 1 year post-treatment) | 267 | 267
Dental Health Assessed 2 Years PT (Eligible, started study treatment, and had dental health assessment 2 years post-treatment) | 208 | 201
Dental Health Assessed 5 Years PT (Eligible, started study treatment, and had dental health assessment 5 years post-treatment) | 44 | 43
Feeding Tube Assessed (Eligible, started study treatment, and had feeding tube assessment 1 year post-treatment) | 368 | 356
Progressed (Eligible and experienced local, regional, or distant progression or death) | 76 | 122
Completed (Subjects contributing any data to analysis are considered to have completed the study) | 406 | 399
Not Completed | 18 | 26
Not completed — Protocol Violation | 17 | 23
Not completed — HIV positive | 1 | 3

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab | Total
Number analyzed (Participants) | 406 | 399 | 805
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [52 to 63] | 58 [52 to 63] | 58 [52 to 63]
Age, Customized [Count of Participants; unit: Participants]
  <= 65 | 344 | 345 | 689
  > 65 | 62 | 54 | 116
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 44 | 77
  Male | 373 | 355 | 728
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 15 | 26
  Not Hispanic or Latino | 383 | 369 | 752
  Unknown or Not Reported | 12 | 15 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 380 | 367 | 747
  Black | 17 | 19 | 36
  Other | 2 | 8 | 10
  Unknown | 7 | 5 | 12
Zubrod performance status [Count of Participants; unit: Participants] — Measure Description: 0 - Asymptomatic; 1 - Symptomatic but completely ambulatory; 2 - Symptomatic, <50% in bed during the day; 3 - Symptomatic, >50% in bed, but not bedbound; 4 - Bedbound; 5 - Death
  Participants
    0 | 295 | 300 | 595
    1 | 111 | 99 | 210
Smoking history [Count of Participants; unit: Participants] — Smoking history as measured in pack-years. It is calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked.
  Participants
    0 pack-years | 194 | 181 | 375
    >0 to <= 10 pack-years | 59 | 68 | 127
    >10 pack-years | 153 | 150 | 303
Smoking history [Median (Inter-Quartile Range); unit: pack-years] — Measure Description: Smoking history as measured in pack-years. It is calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked.
  pack-years | 2 [0 to 22] | 3 [0 to 24] | 2 [0 to 23]
Primary site [Count of Participants; unit: Participants] — Primary location of tumor
  Participants
    Tonsillar fossa, tonsil | 202 | 199 | 401
    Base of tongue | 174 | 179 | 353
    Oropharynx, not otherwise specified | 16 | 15 | 31
    Pharyngeal oropharynx | 8 | 5 | 13
    Soft palate | 4 | 0 | 4
    Vallecula | 2 | 1 | 3
Tumor stage [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 7th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues.
  Participants
    T1 | 89 | 86 | 175
    T2 | 162 | 163 | 325
    T3 | 108 | 100 | 208
    T4 | 47 | 50 | 97
Node category [Count of Participants; unit: Participants] — Regional lymph nodes staging per American Joint Committee on Cancer (AJCC) 7th ed. refers to the number and/or extent of spread of lymph nodes that contain cancer. The higher the number after the N, the greater the involvement of regional lymph nodes.
  Participants
    N0 | 20 | 14 | 34
    N1 | 20 | 25 | 45
    N2a | 59 | 56 | 115
    N2b | 209 | 208 | 417
    N2c | 82 | 83 | 165
    N3 | 16 | 13 | 29
Overall stage [Count of Participants; unit: Participants] — Overall cancer stage per American Joint Committee on Cancer (AJCC) 7th ed. combines tumor (T), regional lymph node (N), and distant metastasis (M) staging to determine an overall stage of 0, I, II, III, or IV, ranging from least to most advanced, respectively. Stage III: T3/N0/M0 or T1-3/N1/M0; Stage IV: T4/any N/M0 or any T/N2-3/M0.
  Participants
    III | 29 | 31 | 60
    IV | 377 | 368 | 745
Risk group per study RTOG-0129 [Count of Participants; unit: Participants] — Risk group as defined by recursive partitioning analysis of study RTOG-0129 (NCT00047008). Low-risk consists of patients with p16-positive tumors and 10 or fewer pack-years or p16-positive, >10 pack-years, and N0-2a disease. Intermediate-risk consists of p16-positive, >10 pack-years, and N2b-3 disease or p16-negative, 10 or fewer pack-years, and T2-3 disease. High-risk consists of p16-negative, 10 or fewer pack-years, and T4 disease or p16-negative and >10 pack-years.
  Participants
    Low risk | 289 | 284 | 573
    Intermediate risk | 117 | 115 | 232

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: An event for overall survival is death due to any cause. Survival time is defined as time from randomization to the date of death or last known follow-up (censored). Rates are estimated by the Kaplan-Meier method. The protocol endpoint is hazard ratio, which is reported in the statistical analysis results. Five-year rate is reported simply as summary data; it is not the outcome measure.
Time Frame: From randomization to last follow-up. Analysis was to occur after 180 deaths were reported. Analysis occurred after 133 deaths were reported. Maximum follow-up at time of analysis was 6.5 years.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 406 | 399
percentage of participants | 84.6 [80.6 to 88.6] | 77.9 [73.4 to 82.5]
Statistical Analysis 1: Comparison: IMRT + Cisplatin vs IMRT + Cetuximab; Test type: Non-Inferiority — The non-inferiority margin was set at 1.45 (hazard ratio scale; IMRT + Cetuximab / IMRT + Cisplatin). If the upper limit of the 95% confidence interval was <1.45, non-inferiority would be concluded. Design was based on a group sequential design with 3 interim analyses, one-sided 0.05, and 80% power; Hazard Ratio (HR) = 1.45, 95% CI 1-sided [upper limit 1.94] — Reference level = IMRT + Cisplatin

2. Secondary Outcome: Progression-free Survival
Description: An event for progression-free survival is local, regional, or distant disease progression or death due to any cause. Progression-free survival time is defined as time from randomization to the date of progression/death or last known follow-up (censored). Rates are estimated by the Kaplan-Meier method. The protocol endpoint is the distribution of progression-free survival times, for which the hazard ratio is reported in the statistical analysis results. Five-year rate is reported simply as summary data; it is not the outcome measure.
Time Frame: as for outcome 1
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 406 | 399
percentage of participants | 78.4 [73.8 to 83.0] | 67.3 [62.4 to 72.2]
Statistical Analysis 1: Comparison: IMRT + Cisplatin vs IMRT + Cetuximab; Test type: Superiority; p = 0.0002, Log Rank; Two-sided significance level = 0.05; Hazard Ratio (HR) = 1.72, 95% CI 2-sided [1.29 to 2.29] — Reference level = IMRT + Cisplatin

3. Secondary Outcome: Time to Local-regional Failure
Description: Failure for local-regional failure endpoint was defined as local or regional progression, salvage surgery of the primary tumor with tumor present/unknown, salvage neck dissection with tumor present/unknown > 20 weeks after the end of radiation therapy, death due to study cancer without documented progression, or death due to unknown causes without documented progression; distant metastasis and death due to other causes were considered competing risks. Local-regional failure time is defined as time from randomization to the date of progression/death or last known follow-up (censored). Rates are estimated by the cumulative incidence method. The protocol endpoint is the distribution of local-regional failure times, for which the hazard ratio is reported in the statistical analysis results. Five-year rate is reported simply as summary data; it is not the outcome measure.
Time Frame: as for outcome 1
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 406 | 399
percentage of participants | 9.9 [6.9 to 13.6] | 17.3 [13.7 to 21.4]
Statistical Analysis 1: Comparison: IMRT + Cisplatin vs IMRT + Cetuximab; Test type: Superiority; p = 0.0005, Log Rank; Two-sided significance level = 0.05; Hazard Ratio (HR) = 2.05, 95% CI 2-sided [1.35 to 3.10] — Reference level = IMRT + Cisplatin

4. Secondary Outcome: Time to Distant Metastasis
Description: Failure for distant metastasis endpoint was defined as distant progression; local-regional failure and death due to any cause were considered competing risks. Distant metastasis time is defined as time from randomization to the date of progression/death or last known follow-up (censored). Rates are estimated by the cumulative incidence method. The protocol endpoint is the distribution of distant metastasis times, for which the hazard ratio is reported in the statistical analysis results. Five-year rate is reported simply as summary data; it is not the outcome measure.
Time Frame: as for outcome 1
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 406 | 399
percentage of participants | 8.6 [5.8 to 11.9] | 11.7 [8.6 to 15.3]
Statistical Analysis 1: Comparison: IMRT + Cisplatin vs IMRT + Cetuximab; Test type: Superiority; p = 0.09, Log Rank — Two-sided significance level = 0.05; Hazard Ratio (HR) = 1.49, 95% CI 2-sided [0.94 to 2.36] — Reference level = IMRT + Cisplatin

5. Secondary Outcome: Time to Secondary Primary Cancer
Description: Failure for second primary endpoint was defined as reporting of a new primary cancer; death due to any cause was considered a competing risk. Second primary time is defined as time from randomization to the date of second primary or last known follow-up (censored). Rates are estimated by the cumulative incidence method. The protocol endpoint is the distribution of second primary cancer times, for which the hazard ratio is reported in the statistical analysis results. Five-year rate is reported simply as summary data; it is not the outcome measure.
Time Frame: as for outcome 1
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 406 | 399
percentage of participants | 9.9 [6.9 to 13.4] | 10.3 [7.1 to 14.2]
Statistical Analysis 1: Comparison: IMRT + Cisplatin vs IMRT + Cetuximab; Test type: Superiority; p = 0.95, Log Rank — Two-sided significance level = 0.05; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.61 to 1.58] — Reference level = IMRT + Cisplatin

6. Secondary Outcome: Distribution of First Progression Events
Description: The first event type for progression-free survival is counted for each participant. Possible first progression events are local, regional, or distant progression, any combination of these, or death. The frequency table of these events is also referred to as "Pattern of failure."
Time Frame: as for outcome 1
Population: Eligible participants with progression-free survival failure
Measure: Count of Participants; unit: Participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 76 | 122
Participants
  Local | 13 | 25
  Regional | 6 | 14
  Local and regional | 4 | 8
  Local and distant | 0 | 1
  Regional and distant | 0 | 5
  Local, regional, and distant | 0 | 2
  Distant | 31 | 43
  Death, due to this disease | 2 | 0
  Death, due to second primary | 1 | 3
  Death, due to other reason | 10 | 11
  Death, due to unknown reason | 9 | 10

7. Secondary Outcome: Percentage of Participants Experiencing Early Death
Description: Early death is defined as death due to adverse event or within 30 days of treatment completion.
Time Frame: as for outcome 1
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 398 | 394
percentage of participants | 1.5 [0.6 to 3.3] | 1.5 [0.6 to 3.3]
Statistical Analysis 1: Comparison: IMRT + Cisplatin vs IMRT + Cetuximab; Test type: Superiority; p = 1.0, Fisher Exact — Two-sided significance level = 0.05

8. Secondary Outcome: Percentage of Participants With Acute Grade 3-4 Treatment-related Adverse Events: During Treatment
Description: Acute adverse events (AE) are defined as occurring within 180 days from the end of treatment. "Treatment-related" means reported as definitely, probably, or possibly related to protocol treatment. AE were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Grade refers to the severity of the AE. The CTCAE v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to AE
Time Frame: From start of treatment to end of treatment, approximately 6 weeks
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 398 | 394
percentage of participants | 75.6 [71.1 to 79.8] | 73.6 [69.0 to 77.9]

9. Secondary Outcome: Percentage of Participants With Acute Grade 3-4 Treatment-related Adverse Events: 1 Month After End of Study Treatment
Description: as for outcome 8
Time Frame: From start of treatment to approximately 2.5 months (1 month after the end of treatment)
Population: Eligible patients who started study treatment and had adverse events assessment at 1 month after treatment end
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 369 | 363
percentage of participants | 32.5 [27.8 to 37.6] | 31.1 [26.4 to 36.2]

10. Secondary Outcome: Percentage of Participants With Acute Grade 3-4 Treatment-related Adverse Events: 3 Months After the End of Study Treatment
Description: as for outcome 8
Time Frame: From start of treatment to approximately 4.5 months (3 months after the end of treatment)
Population: Eligible patients who started study treatment and had adverse events assessment at 3 months after treatment end
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 359 | 367
percentage of participants | 17.5 [13.8 to 21.9] | 14.7 [11.3 to 18.8]

11. Secondary Outcome: Percentage of Participants With Acute Grade 3-4 Treatment-related Adverse Events: 6 Months After the End of Study Treatment
Description: as for outcome 8
Time Frame: From start of treatment to approximately 7.5 months (6 months after the end of treatment)
Population: Eligible patients who started study treatment and had adverse events assessment at 6 months year after treatment end
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 361 | 352
percentage of participants | 13.3 [10.0 to 17.2] | 9.4 [6.5 to 12.9]

12. Secondary Outcome: Percentage of Participants With Late Grade 3-4 Treatment-related Adverse Events: 1 Year After the End of Study Treatment
Description: Late adverse events (AE) are defined as > 180 days from end of treatment. "Treatment-related" means reported as definitely, probably, or possibly related to protocol treatment. AE were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Grade refers to the severity of the AE. The CTCAE v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to AE
Time Frame: From start of treatment to approximately 13.5 months (one year after the end of treatment)
Population: Eligible patients who started study treatment and had adverse events assessment at 1 year after treatment end
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 360 | 351
percentage of participants | 10.0 [7.1 to 13.6] | 8.5 [5.8 to 12.0]

13. Secondary Outcome: Percentage of Participants With Late Grade 3-4 Treatment-related Adverse Events: 2 Years After the End of Study Treatment
Description: as for outcome 12
Time Frame: From 180 days after end of treatment to two years after end of treatment.
Population: .Eligible patients who started study treatment and had adverse events assessment at 2 years after treatment end
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 311 | 303
percentage of participants | 7.7 [5.0 to 11.3] | 4.0 [2.1 to 6.8]

14. Secondary Outcome: Percentage of Participants With Late Grade 3-4 Treatment-related Adverse Events: 5 Years After the End of Study Treatment
Description: as for outcome 12
Time Frame: From start of treatment to approximately 61.5 months (five years after the end of treatment)
Population: Eligible patients who started study treatment and had adverse events assessment at 5 years after treatment end
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 92 | 86
percentage of participants | 4.3 [1.2 to 10.8] | 7.0 [2.6 to 14.6]

15. Secondary Outcome: Percentage of Participants With a Feeding Tube at 1 Year
Time Frame: From randomization to 1 year.
Population: Eligible patients who started study treatment and had feeding tube assessment at 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 368 | 356
percentage of participants | 9.2 [6.5 to 12.7] | 8.4 [5.8 to 11.8]
Statistical Analysis 1: Comparison: IMRT + Cisplatin; Test type: Superiority; p = 0.79, Fisher Exact — Two-sided significance level = 0.05

16. Secondary Outcome: EORTC QLQ-C30 Global Health Status Score Change From Baseline at End of Treatment
Description: The EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30) Global Health Status score measures a cancer patient's perception of their overall health and well-being and ranges from 0 (worst) to 100 (best). A positive change from baseline indicates improvement.
Time Frame: Baseline and end of treatment (6-7 weeks)
Population: Eligible participants enrolled to the quality of life (QOL) substudy who received protocol treatment and had outcome measure data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 131 | 133
score on a scale | -23.16 (28.16) | -25.31 (22.92)

17. Secondary Outcome: EORTC QLQ-C30 Global Health Status Score Change From Baseline at 3 Months From End of Treatment
Description: The EORTC QLQ-C30 Global Health Status score measures a cancer patient's perception of their overall health and well-being and ranges from 0 (worst) to 100 (best). A positive change from baseline indicates improvement.
Time Frame: Baseline and 3 months from end of treatment. Treatment lasts 6-7 weeks.
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 130 | 132
score on a scale | -4.42 (25.92) | -7.51 (22.46)

18. Secondary Outcome: EORTC QLQ-C30 Global Health Status Score Change From Baseline at 6 Months From End of Treatment
Description: as for outcome 17
Time Frame: Baseline and 6 months from end of treatment. Treatment lasts 6-7 weeks.
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 132 | 130
score on a scale | -0.57 (25.01) | -0.90 (23.35)
Statistical Analysis 1: Comparison: IMRT + Cisplatin vs IMRT + Cetuximab; Test type: Superiority; p = 0.5438, t-test, 1 sided — One-sided significance level = 0.05

19. Secondary Outcome: EORTC QLQ-C30 Global Health Status Score Change From Baseline at 12 Months From End of Treatment
Description: as for outcome 17
Time Frame: Baseline and 12 months from end of treatment. Treatment lasts 6-7 weeks
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 119 | 116
score on a scale | 3.15 (23.42) | 2.59 (21.09)

20. Secondary Outcome: EORTC QLQ-H&N35 Swallowing Score Change From Baseline at End of Treatment
Description: The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Head and Neck Cancer Module (EORTC QLQ-H&N35) swallowing score measures patient-reported difficulty with swallowing various foods and liquid and ranges from 0 (no swallowing problems) to 100 (maximum swallowing difficulty). A positive change from baseline indicates worsening swallowing function.
Time Frame: Baseline and end of treatment (6-7 weeks)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 131 | 132
score on a scale | 47.99 (27.99) | 47.43 (24.52)

21. Secondary Outcome: EORTC QLQ-H&N35 Swallowing Score Change From Baseline at 3 Months From End of Treatment.
Description: The EORTC QLQ-H&N35 swallowing score measures patient-reported difficulty with swallowing various foods and liquid and ranges from 0 (no swallowing problems) to 100 (maximum swallowing difficulty). A positive change from baseline indicates worsening swallowing function.
Time Frame: Baseline and 3 months from end of treatment. Treatment lasts 6-7 weeks.
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 130 | 132
score on a scale | 10.58 (26.49) | 14.20 (20.61)

22. Secondary Outcome: EORTC QLQ-H&N35 Swallowing Score Change From Baseline at 6 Months From End of Treatment.
Description: as for outcome 21
Time Frame: Baseline and 6 months from end of treatment. Treatment lasts 6-7 weeks.
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 132 | 130
score on a scale | 8.65 (23.94) | 10.13 (18.73)
Statistical Analysis 1: Comparison: IMRT + Cisplatin vs IMRT + Cetuximab; Test type: Superiority; p = 0.7108, t-test, 1 sided — One-sided significance level = 0.05

23. Secondary Outcome: EORTC QLQ-H&N35 Swallowing Score Change From Baseline at 12 Months From End of Treatment.
Description: as for outcome 21
Time Frame: Baseline and 12 months from end of treatment. Treatment lasts 6-7 weeks.
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 119 | 116
score on a scale | 2.52 (19.64) | 7.61 (17.81)

24. Secondary Outcome: Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events for Head and Neck (PRO-CTCAE H&N) at Baseline, End of Treatment, 3, 6, and 12 Months From End of Treatment.
Time Frame: From randomization to 1 year after end of treatment.
Reporting Status: Not Posted, anticipated posting 2026-06

25. Secondary Outcome: EuroQol Five Dimension Scale (EQ-5D) at Baseline, End of Treatment, 3, 6, and 12 Months From End of Treatment.
Time Frame: From randomization to 1 year after end of treatment.
Reporting Status: Not Posted, anticipated posting 2026-06

26. Secondary Outcome: Work Status Questionnaire at Baseline, End of Treatment, 3, 6, and 12 Months.
Time Frame: From randomization to 1 year after end of treatment.
Reporting Status: Not Posted, anticipated posting 2026-06

27. Secondary Outcome: Percentage of Patients With Normal/Good Dental Health: Pretreatment
Description: This study utilized a dental effects health scale from 0 (normal) to 4 (life-threatening dental condition). The percentage of participants with a value of 0 or 1 is reported: 0 = "Normal: Edentulous, with no gingival disease";
  1 = "Mild changes/good dental health: mild periodontal inflammation-routine cleaning indicated; < 5 restorations indicated; no extractions indicated." Ten year data is not yet available.
Time Frame: Before treatment
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 398 | 394
percentage of participants | 71.1 [66.4 to 75.5] | 74.6 [70.0 to 78.8]

28. Secondary Outcome: Percentage of Patients With Normal/Good Dental Health: 1 Year After End of Treatment
Description: This study utilized a dental effects health scale from 0 (normal) to 4 (life-threatening dental condition). The percentage of participants with a value of 0 or 1 is reported: 0 = "Normal: Edentulous, with no gingival disease";
  1 = "Mild changes/good dental health: mild periodontal inflammation-routine cleaning indicated; < 5 restorations indicated; no extractions indicated."
Time Frame: 1 year after end of treatment (approximately 13.5 months)
Population: Eligible patients who started study treatment and had dental status assessment at 1 year after treatment end
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 267 | 267
percentage of participants | 87.3 [82.7 to 91.0] | 83.5 [78.5 to 87.8]

29. Secondary Outcome: Percentage of Patients With Normal/Good Dental Health: 2 Years After End of Treatment
Description: as for outcome 28
Time Frame: 2 years after end of treatment (approximately 25.5 months)
Population: Eligible patients who started study treatment and had dental status assessment at 2 years after treatment end
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 208 | 201
percentage of participants | 86.5 [81.1 to 90.9] | 82.1 [76.1 to 87.1]

30. Secondary Outcome: Percentage of Patients With Normal/Good Dental Health: 5 Years After End of Treatment
Description: as for outcome 28
Time Frame: 5 years after end of treatment (approximately 61.5 months)
Population: Eligible patients who started study treatment and had dental status assessment at 5 years after treatment end
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 44 | 43
percentage of participants | 88.6 [75.4 to 96.2] | 86.0 [72.1 to 94.7]

31. Secondary Outcome: Percentage of Patients With Normal/Good Dental Health: 10 Years After End of Treatment
Description: as for outcome 28
Time Frame: 10 years after end of treatment (approximately 121.5 months)
Population: Eligible patients who started study treatment and had dental status assessment at 10 years after treatment end
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 34 | 25
Percentage of participants | 91.2 [76.3 to 98.1] | 84.0 [63.9 to 95.5]

32. Secondary Outcome: Number of Participants by HHIA-S Category at Baseline
Description: The Hearing Handicap Inventory for Adults Screen Version (HHIA-S) measures a person's perceived hearing handicap. Total score ranges from 0 to 40, with a higher score indicating more severe perceived hearing handicap, categorized as follows:
  * No handicap: 0-8.
  * Mild-moderate handicap: 10-24.
  * Severe handicap: 26-40.
Time Frame: Baseline
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 175 | 171
Participants
  No handicap | 150 | 132
  Mild-moderate handicap | 23 | 32
  Severe handicap | 2 | 7

33. Secondary Outcome: Number of Participants by HHIA-S Category at End of Treatment
Description: as for outcome 32
Time Frame: End of treatment (6-7 weeks)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 134 | 133
Participants
  No handicap | 91 | 107
  Mild-moderate handicap | 29 | 21
  Severe handicap | 14 | 5

34. Secondary Outcome: Number of Participants by HHIA-S Category at 3 Months After End of Treatment
Description: The HHIA-S measures a person's perceived hearing handicap. Total score ranges from 0 to 40, with a higher score indicating more severe perceived hearing handicap, categorized as follows:
  * No handicap: 0-8.
  * Mild-moderate handicap: 10-24.
  * Severe handicap: 26-40.
Time Frame: 3 months after end of treatment. Treatment lasts 6-7 weeks.
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 136 | 137
Participants
  No handicap | 93 | 109
  Mild-moderate handicap | 28 | 21
  Severe handicap | 15 | 7

35. Secondary Outcome: Number of Participants by HHIA-S Category at 6 Months After End of Treatment
Description: as for outcome 34
Time Frame: 6 months after end of treatment. Treatment lasts 6-7 weeks.
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 140 | 131
Participants
  No handicap | 95 | 106
  Mild-moderate handicap | 31 | 21
  Severe handicap | 14 | 4

36. Secondary Outcome: Number of Participants by HHIA-S Category at 12 Months After End of Treatment
Description: as for outcome 34
Time Frame: 12 months after end of treatment. Treatment lasts 6-7 weeks.
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 121 | 125
Participants
  No handicap | 84 | 103
  Mild-moderate handicap | 27 | 17
  Severe handicap | 10 | 5

37. Secondary Outcome: Overall Survival by KRAS (Kirsten Rat Sarcoma Viral Oncogene Homolog) Variant Status
Description: KRAS (Kirsten Rat Sarcoma Viral Oncogene Homolog) is a gene that helps control how cells grow. Some people have a change in this gene, which can be detected (variant/non-variant) by a genetic test performed on tissue from their tumor. Research suggests that this change may influence how head and neck cancer responds to certain treatments.
  An event for overall survival is death due to any cause. Survival time is defined as time from randomization to the date of death or last known follow-up (censored). Rates are estimated by the Kaplan-Meier method. The protocol endpoint is hazard ratio, which is reported in the statistical analysis results. Five-year rate is reported simply as summary data; it is not the outcome measure.
Time Frame: From randomization to last follow-up. Analysis was to occur after 180 deaths were reported. Analysis occurred after 214 deaths were reported. Median follow-up at time of analysis was 8.3 years.
Population: Eligible participants with KRAS data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Variant: Has the KRAS variant
- Non-variant: Does not have the KRAS variant
Arm/Group | Variant | Non-variant
Number analyzed (Participants) | 92 | 470
percentage of participants | 80.6 [72.3 to 88.9] | 79.2 [75.4 to 83.0]
Statistical Analysis 1: Comparison: Variant vs Non-variant; Test type: Superiority; p = 0.2571, Regression, Cox — One-sided significance level = 0.025; Stratified by treatment arm; Cox Proportional Hazard = 0.87, 95% CI 2-sided [0.56 to 1.34] — Reference level = non-variant

38. Secondary Outcome: Progression-free Survival by KRAS Variant Status
Description: KRAS (Kirsten Rat Sarcoma Viral Oncogene Homolog) is a gene that helps control how cells grow. Some people have a change in this gene, which can be detected (variant/non-variant) by a genetic test performed on tissue from their tumor. Research suggests that this change may influence how head and neck cancer responds to certain treatments.
  An event for progression-free survival is local, regional, or distant disease progression or death due to any cause. Progression-free survival time is defined as time from randomization to the date of progression/death or last known follow-up (censored). Rates are estimated by the Kaplan-Meier method. The protocol endpoint is the distribution of progression-free survival times, for which the hazard ratio is reported in the statistical analysis results. Five-year rate is reported simply as summary data; it is not the outcome measure.
Time Frame: as for outcome 37
Population: Eligible participants with KRAS data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Variant | Non-variant
Number analyzed (Participants) | 92 | 470
percentage of participants | 72.0 [62.6 to 81.3] | 71.5 [67.3 to 75.7]
Statistical Analysis 1: Comparison: Variant vs Non-variant; Test type: Superiority; p = 0.3704, Regression, Cox — One-sided significance level = 0.05; Stratified by treatment arm; Cox Proportional Hazard = 0.94, 95% CI 2-sided [0.64 to 1.38] — Reference level = non-variant

39. Secondary Outcome: Overall Survival by Treatment Arm Within KRAS Variant Status Group
Description: as for outcome 37
Time Frame: as for outcome 37
Population: Eligible participants with KRAS data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 275 | 287
percentage of participants
  Variant: number analyzed (Participants) | 44 | 48
  Variant | 83.3 [72.0 to 94.6] | 78.4 [66.5 to 90.3]
  Non-variant: number analyzed (Participants) | 231 | 239
  Non-variant | 80.8 [75.6 to 86.1] | 77.6 [72.2 to 83.1]
Statistical Analysis 1: Comparison: IMRT + Cisplatin vs IMRT + Cetuximab; Variant; Test type: Superiority; Cox Proportional Hazard = 1.10, 95% CI 2-sided [0.49 to 2.46] — Reference level = IMRT + Cisplatin
Statistical Analysis 2: Comparison: IMRT + Cisplatin vs IMRT + Cetuximab; Non-variant; Test type: Superiority; Cox Proportional Hazard = 1.10, 95% CI [0.79 to 1.53] — Reference level = IMRT + Cisplatin
Statistical Analysis 3: Comparison: IMRT + Cisplatin vs IMRT + Cetuximab; Testing Cox proportional hazards model interaction term for KRAS variant status and treatment arm; Test type: Other; p = 0.9890, Regression, Cox — Two-sided significance level = 0.05

40. Secondary Outcome: Progression-free Survival Within KRAS Variant Status
Description: as for outcome 38
Time Frame: as for outcome 37
Population: Eligible participants with KRAS data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 275 | 287
percentage of participants
  Variant: number analyzed (Participants) | 44 | 48
  Variant | 76.6 [63.9 to 89.3] | 67.7 [54.2 to 81.2]
  Non-variant: number analyzed (Participants) | 231 | 239
  Non-variant | 75.1 [69.4 to 80.8] | 68.0 [62.0 to 74.1]
Statistical Analysis 1: Comparison: IMRT + Cisplatin vs IMRT + Cetuximab; Variant; Test type: Superiority; Cox Proportional Hazard = 1.01, 95% CI [0.50 to 2.04] — Reference level = IMRT + Cisplatin
Statistical Analysis 2: Comparison: IMRT + Cisplatin vs IMRT + Cetuximab; Non-variant; Test type: Superiority; Cox Proportional Hazard = 1.27, 95% CI 2-sided [0.94 to 1.73] — Reference level = IMRT + Cisplatin
Statistical Analysis 3: Comparison: IMRT + Cisplatin vs IMRT + Cetuximab; Testing Cox proportional hazards model interaction term for KRAS variant status and treatment arm; Test type: Other; p = 0.5556, Regression, Cox — Two-sided significance level = 0.05

41. Other Pre Specified Outcome: Overall Survival by Sex
Description: NIH-required analysis. An event for overall survival is death due to any cause. Survival time is defined as time from randomization to the date of death or last known follow-up (censored). Rates are estimated by the Kaplan-Meier method. The protocol endpoint is hazard ratio, which is reported in the statistical analysis results. Five-year rate is reported simply as summary data; it is not the outcome measure.
Time Frame: as for outcome 1
Population: Eligible participants. Data were stratified by sex.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 406 | 399
percentage of participants
  Female: number analyzed (Participants) | 33 | 44
  Female | 93.4 [84.6 to 100] | 76.8 [62.8 to 90.8]
  Male: number analyzed (Participants) | 373 | 355
  Male | 83.8 [79.6 to 88.1] | 78.0 [73.2 to 82.9]

42. Other Pre Specified Outcome: Overall Survival by Ethnicity
Description: as for outcome 41
Time Frame: as for outcome 1
Population: Eligible participants. Data were stratified by ethnicity.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 406 | 399
percentage of participants
  Hispanic or Latino: number analyzed (Participants) | 11 | 15
  Hispanic or Latino | 100 [NA to NA] — SAS software does not compute a confidence interval when the estimate is 100%. | 70.7 [46.5 to 95.0]
  Not Hispanic or Latino: number analyzed (Participants) | 383 | 369
  Not Hispanic or Latino | 84.7 [80.6 to 88.8] | 77.9 [73.2 to 82.7]
  Unknown or Not Reported: number analyzed (Participants) | 12 | 15
  Unknown or Not Reported | 66.8 [35.1 to 98.6] | 85.7 [67.4 to 100]

43. Other Pre Specified Outcome: Overall Survival by Race
Description: as for outcome 41
Time Frame: From randomization to last follow-up. Analysis was to occur after 180 deaths were reported. Analysis occurred after 133 deaths were reported. Maximum follow-up at time of analysis was 6.5 years. Five-year rates are reported here.
Population: Eligible participants. Data were stratified by ethnicity.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
Number analyzed (Participants) | 406 | 399
percentage of participants
  American Indian or Alaska Native: number analyzed (Participants) | 0 | 2
  American Indian or Alaska Native |  | 100 [NA to NA] — SAS software does not compute a confidence interval when the estimate is 100%.
  Asian: number analyzed (Participants) | 2 | 1
  Asian | NA [NA to NA] — Cannot be calculated because participants was censored prior to the timepoint. | 100 [NA to NA] — SAS software does not compute a confidence interval when the estimate is 100%
  Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 0 | 2
  Native Hawaiian or Other Pacific Islander |  | NA [NA to NA] — Cannot be calculated because participants were censored prior to the timepoint.
  Black or African American: number analyzed (Participants) | 17 | 19
  Black or African American | 77.5 [54.9 to 100] | 76.4 [55.9 to 96.9]
  White: number analyzed (Participants) | 380 | 367
  White | 84.6 [80.5 to 88.7] | 77.3 [72.5 to 82.1]
  More than one race: number analyzed (Participants) | 0 | 3
  More than one race |  | NA [NA to NA] — Cannot be calculated because participants were censored prior to the timepoint.
  Unknown or Not Reported: number analyzed (Participants) | 7 | 5
  Unknown or Not Reported | 100 [NA to NA] — SAS software does not compute a confidence interval when the estimate is 100%. | 100 [NA to NA] — SAS software does not compute a confidence interval when the estimate is 100%.

ADVERSE EVENTS:
Time Frame: From randomization to last follow-up. Maximum follow-up was 7.4 years.
Description: Eligible patients who started treatment are included. Patients experiencing more than one of a given adverse event are counted only once for that adverse event
Arm/Group | IMRT + Cisplatin | IMRT + Cetuximab
All-Cause Mortality (participants affected / at risk) | 64/406 | 86/399
Serious Adverse Events (participants affected / at risk) | 177/398 | 115/394
Other Adverse Events (participants affected / at risk) | 398/398 | 393/394
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT + Cisplatin (N=398) | IMRT + Cetuximab (N=394)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 14 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Spleen disorder (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Aortic valve disease (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 2
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardiac disorders - Other (Cardiac disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 2
Sinus tachycardia (Cardiac disorders) | 2 | 3
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 3 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Colonic fistula (Gastrointestinal disorders) | 1 | 0
Colonic perforation (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 11 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 23 | 17
Esophageal pain (Gastrointestinal disorders) | 2 | 1
Esophageal stenosis (Gastrointestinal disorders) | 3 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 4
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 18 | 22
Nausea (Gastrointestinal disorders) | 38 | 18
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Oral cavity fistula (Gastrointestinal disorders) | 1 | 0
Oral hemorrhage (Gastrointestinal disorders) | 1 | 1
Oral pain (Gastrointestinal disorders) | 7 | 2
Pancreatitis (Gastrointestinal disorders) | 2 | 1
Rectal pain (Gastrointestinal disorders) | 0 | 1
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 34 | 14
Death NOS (General disorders) | 0 | 1
Fatigue (General disorders) | 6 | 3
Fever (General disorders) | 8 | 8
Flu like symptoms (General disorders) | 1 | 0
Infusion related reaction (General disorders) | 0 | 8
Localized edema (General disorders) | 1 | 0
Pain (General disorders) | 12 | 9
Sudden death NOS (General disorders) | 4 | 2
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 0 | 1
Anaphylaxis (Immune system disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Anorectal infection (Infections and infestations) | 1 | 1
Bronchial infection (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 2 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 2
Infections and infestations - Other (Infections and infestations) | 2 | 2
Joint infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 7 | 5
Mucosal infection (Infections and infestations) | 3 | 1
Rash pustular (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 1
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 2 | 2
Soft tissue infection (Infections and infestations) | 2 | 1
Upper respiratory infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 5
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 1
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 2 | 2
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
CPK increased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 5 | 0
INR increased (Investigations) | 1 | 0
Investigations - Other (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 12 | 11
Neutrophil count decreased (Investigations) | 13 | 0
Weight gain (Investigations) | 1 | 0
Weight loss (Investigations) | 8 | 5
White blood cell decreased (Investigations) | 6 | 0
Anorexia (Metabolism and nutrition disorders) | 9 | 4
Dehydration (Metabolism and nutrition disorders) | 43 | 20
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 8 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 4 | 4
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Movements involuntary (Nervous system disorders) | 0 | 1
Myelitis (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 6 | 1
Transient ischemic attacks (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Confusion (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Hallucinations (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 21 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pharyngeal necrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 3 | 0
Lymphedema (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 8 | 2
Vascular disorders - Other (Vascular disorders) | 3 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT + Cisplatin (N=398) | IMRT + Cetuximab (N=394)
Anemia (Blood and lymphatic system disorders) | 185 | 118
Ear pain (Ear and labyrinth disorders) | 30 | 36
Hearing impaired (Ear and labyrinth disorders) | 192 | 104
Tinnitus (Ear and labyrinth disorders) | 204 | 100
Hyperthyroidism (Endocrine disorders) | 20 | 10
Hypothyroidism (Endocrine disorders) | 74 | 69
Abdominal pain (Gastrointestinal disorders) | 21 | 15
Constipation (Gastrointestinal disorders) | 240 | 214
Diarrhea (Gastrointestinal disorders) | 94 | 87
Dry mouth (Gastrointestinal disorders) | 376 | 372
Dyspepsia (Gastrointestinal disorders) | 123 | 88
Dysphagia (Gastrointestinal disorders) | 371 | 351
Gastroesophageal reflux disease (Gastrointestinal disorders) | 13 | 23
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 54 | 61
Mucositis oral (Gastrointestinal disorders) | 363 | 370
Nausea (Gastrointestinal disorders) | 301 | 238
Oral pain (Gastrointestinal disorders) | 34 | 60
Salivary duct inflammation (Gastrointestinal disorders) | 32 | 34
Vomiting (Gastrointestinal disorders) | 206 | 150
Chills (General disorders) | 19 | 27
Fatigue (General disorders) | 357 | 345
Fever (General disorders) | 22 | 46
General disorders and administration site conditions - Other (General disorders) | 11 | 20
Neck edema (General disorders) | 42 | 33
Pain (General disorders) | 329 | 324
Infections and infestations - Other (Infections and infestations) | 29 | 32
Mucosal infection (Infections and infestations) | 53 | 43
Dermatitis radiation (Injury, poisoning and procedural complications) | 316 | 305
Alanine aminotransferase increased (Investigations) | 52 | 67
Alkaline phosphatase increased (Investigations) | 18 | 20
Aspartate aminotransferase increased (Investigations) | 35 | 53
Creatinine increased (Investigations) | 97 | 23
Investigations - Other (Investigations) | 21 | 14
Lymphocyte count decreased (Investigations) | 98 | 101
Neutrophil count decreased (Investigations) | 106 | 17
Platelet count decreased (Investigations) | 100 | 23
Weight loss (Investigations) | 203 | 211
White blood cell decreased (Investigations) | 157 | 53
Anorexia (Metabolism and nutrition disorders) | 263 | 253
Dehydration (Metabolism and nutrition disorders) | 97 | 68
Hyperglycemia (Metabolism and nutrition disorders) | 90 | 97
Hyperkalemia (Metabolism and nutrition disorders) | 25 | 17
Hypermagnesemia (Metabolism and nutrition disorders) | 20 | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 94 | 101
Hypocalcemia (Metabolism and nutrition disorders) | 73 | 45
Hypokalemia (Metabolism and nutrition disorders) | 64 | 48
Hypomagnesemia (Metabolism and nutrition disorders) | 64 | 66
Hyponatremia (Metabolism and nutrition disorders) | 132 | 81
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 21 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 16
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 32 | 29
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 38 | 31
Neck pain (Musculoskeletal and connective tissue disorders) | 46 | 44
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 21 | 20
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 29 | 48
Trismus (Musculoskeletal and connective tissue disorders) | 98 | 103
Dizziness (Nervous system disorders) | 51 | 33
Dysgeusia (Nervous system disorders) | 349 | 334
Headache (Nervous system disorders) | 47 | 65
Peripheral sensory neuropathy (Nervous system disorders) | 104 | 62
Anxiety (Psychiatric disorders) | 45 | 60
Depression (Psychiatric disorders) | 49 | 44
Insomnia (Psychiatric disorders) | 135 | 118
Cough (Respiratory, thoracic and mediastinal disorders) | 147 | 127
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 33 | 30
Hiccups (Respiratory, thoracic and mediastinal disorders) | 35 | 10
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 83 | 81
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 13 | 23
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 137 | 116
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 13 | 25
Sore throat (Respiratory, thoracic and mediastinal disorders) | 71 | 65
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 30 | 34
Alopecia (Skin and subcutaneous tissue disorders) | 111 | 89
Dry skin (Skin and subcutaneous tissue disorders) | 106 | 140
Pruritus (Skin and subcutaneous tissue disorders) | 42 | 105
Rash acneiform (Skin and subcutaneous tissue disorders) | 21 | 300
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 28 | 96
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 30 | 48
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 41 | 49
Telangiectasia (Skin and subcutaneous tissue disorders) | 24 | 18
Hypertension (Vascular disorders) | 43 | 39
Hypotension (Vascular disorders) | 24 | 17
Lymphedema (Vascular disorders) | 32 | 37

LIMITATIONS AND CAVEATS:
At the third interim analysis the NRG Oncology Data Monitoring Committee recommended the public release of study results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-02-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT01302834/Prot_SAP_001.pdf
  • Informed Consent Form (2016-02-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT01302834/ICF_000.pdf